CLINICAL TRIAL: NCT02654496
Title: The Gut Microbiota in Patients Post Roux-en-Y Gastric Bypass Surgery
Brief Title: Gut Microbiota Post Roux-en-Y Gastric Bypass Surgery
Status: Completed | Type: Observational
Sponsor: North Dakota State University (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University
Other Study IDs: IRB-201509-061
Record Dates: First submitted 2015-12-17; First posted 2016-01-13 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Gut Microbiota; Weight Regain; Gastric Bypass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Fecal Samples and Plasma/Serum Samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1 (Successful weight loss): 3-5 years post Roux-en-Y gastric bypass patients who had successful weight loss
  Interventions: Other: Meal challenge
- Group 2 (Suboptimal weight loss): 3-5 years post Roux-en-Y gastric bypass patients who had suboptimal weight loss
  Interventions: Other: Meal challenge
- Group 3 (Control group): A control group who has not had Roux-en-Y gastric bypass surgery and are of similar age, gender, body mass index as the gastric bypass groups.
  Interventions: Other: Meal challenge

INTERVENTIONS:
Other: Meal challenge — Participants will receive a liquid nutritional supplement. Before and after administration, biological variables of interest will be collected.

SUMMARY:
The purpose of this study is to investigate mechanisms responsible for weight change in patients who have undergone weight loss surgery. Specifically, we will compare the gut microbiota, plasma bile acids, plasma gut peptides (GLP-1, GLP-2, and PYY), and plasma LPS in three groups of subjects: 3-5 years post gastric bypass patients who experienced sub-optimal weight loss, 3-5 years post gastric bypass patients who had successful weight loss, and a control group who has not had a weight loss surgery and are of similar age, gender, body mass index as the gastric bypass groups.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-65
* 3-5 years post Roux-en-Y gastric bypass and experienced successful weight loss following surgery (up to n=10) or
* 3-5 years post Roux-en-Y gastric bypass and did not experience optimal weight loss following surgery (up to n=10) or
* Nonsurgical control participants who are approximately matched in sex, age, and BMI to the optimal weight loss group (up to n=10).

Exclusion Criteria:

* Tobacco use in past three months.
* Taking a medication which is known to significantly influence gastrointestinal transit time or affect the microbiome or other variables significantly (as determined by study pharmacist/MD).
* History of diabetes mellitus.
* Has taken an oral or IV/IM antibiotic in the past 3 months.
* Has taken probiotic and/or prebiotic agent in the past 3 months
* History of significant intestinal disease or disorder (e.g., Crohn's disease, ulcerative colitis, irritable bowel syndrome)
* History of gastrointestinal surgery that may impact measures of biological variables, as determined by the investigator.
* Medical condition expected to impact the biological variables of interest or interfere with providing a sample, as determined by the investigator.
* Unable to speak/read English.
* Breastfeeding, pregnant, or planning to become pregnant within the duration of the study.
* Unwilling to use a medically acceptable form of contraception.
* History of bipolar or psychotic spectrum disorder or alcohol or substance treatment in the past year

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3-5 years post gastric bypass patients and control subjects
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Intestinal Microbiome Composition. The ratio of firmicutes to bacteroidetes will be the primary focus of the microbiome evaluation. | 3-5 years post RYGB

SECONDARY OUTCOMES:
Plasma levels of cholic acid, chenodeoxy cholic acids, deoxycholic acid, and lithocholic acid will be measured by LCMS and will be compared between successful weight loss and poor weight loss post-RYGB and control groups. | 3-5 years post RYGB
Plasma levels of GLP-1, GLP-2, and PYY will be measured by ELISA and will be compared between successful weight loss and poor weight loss post-RYGB and control groups. | 3-5 years post RYGB
Plasma levels of Lipopolysaccharide (LPS) will be measured by the Limulus Amebocyte Lysate (LAL) assay and will be compared between successful weight loss and poor weigh loss post-RYGB and control groups. | 3-5 years post RYGB

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Steffen, PharmD.,Ph.D, Principal Investigator — North Dakota State University
Locations (1):
- North Dakota State University/Sanford Health, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Derived] Fouladi F, Brooks AE, Fodor AA, Carroll IM, Bulik-Sullivan EC, Tsilimigras MCB, Sioda M, Steffen KJ. The Role of the Gut Microbiota in Sustained Weight Loss Following Roux-en-Y Gastric Bypass Surgery. Obes Surg. 2019 Apr;29(4):1259-1267. doi: 10.1007/s11695-018-03653-y. PMID 30604078